CLINICAL TRIAL: NCT07038720
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, and Food Effect of UA026 Tablets in Healthy Adult Subjects and Adult Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study of UA026 Tablets in Healthy Adult Subjects and Adult Subjects With Moderate to Severe Plaque Psoriasis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Usynova Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UA026-CN101
Record Dates: First submitted 2025-06-08; First posted 2025-06-26 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Plaque Psoriasis; Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UA026 (Experimental): Part A: SAD in healthy subjects
  Part B: MAD in healthy subjects
  Part C: FE in healthy subjects
  Part D: Multiple dose study in psoriasis patients
  Interventions: Drug: UA026
- Placebo (Placebo Comparator): Part A: SAD in healthy subjects
  Part B: MAD in healthy subjects
  Part D: Multiple dose study in psoriasis patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UA026 — UA026 will be administered as tablet
  Arms: UA026
Drug: Placebo — Matching placebo will be administered as tablet
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetic profile, and food effect of UA026 tablets.

The study consists of four parts: Part A is a single ascending dose (SAD) study, Part B is a multiple ascending dose (MAD) study, Part C is a food effect (FE) study, and Part D is a multi-dose parallel control study. Part A, B, and C will be conducted in healthy subject, and Part D will be conducted in subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
Interleukin (IL)-17A is a proinflammatory cytokine that when dysregulated can lead to inflammatory disorders. Inhibiting IL-17A has shown remarkable clinical efficacy in psoriasis.UA026 is a high potency small molecule IL-17A inhibitor. This first-in-human study assessed the safety, tolerability, pharmacokinetics (PKs), and biomarkers including circulating IL-17A target engagement profile of single or multiple oral doses of the UA026 in healthy subject and subjects with moderate to severe plaque psoriasis.

ELIGIBILITY:
For Healthy Subject:

Inclusion Criteria

1. Men and women aged 18-55 at the time of screening visit;
2. Body mass index (BMI) 18.5-28 kg/m2, inclusive, and total body weight ≥50 kg for male or ≥45 kg for female;
3. Voluntarily participate in the study and provide the signed and dated informed consent;
4. For female subjects:

   1. With no childbearing potential, including those who has surgical sterilization (documented tubal ligation, hysterectomy, or bilateral oophorectomy) at least 6 weeks before the screening visit, and who menopause ≥12 months before the screening visit (confirmed by a follicle stimulating hormone (FSH) level ≥40IU/L), or
   2. With childbearing potential (WOCBP), must not be pregnant nor lactating, and must have used nonpharmacologic contraception 30 days before administration, during the study, and for 3 months after dose, and must have tested negative for human chorionic gonadotropin (hCG) at the screening visit and D-1; female subjects must refrain from egg donation during this period.
5. Males who are sexually active with WOCBP must have used nonpharmacologic contraception 14 days before administration, during the study, and for 3 months after administration. Male subjects must refrain from sperm donation during this time.
6. Subject is willing to comply with protocol-specified visits, treatments, laboratory tests, and other study-related procedures and requirements.

Exclusion Criteria

1. Allergy to the investigational drugs or the excipients, or a history of severe allergy (including any food allergy or drug allergy);
2. Has received IL-17 small molecule inhibitors in the past;
3. Medical history or family history of psychiatric disorders or genetic immunodeficiency;
4. Has received hematopoietic stem cell transplantation, or organ transplantation in the past;
5. History of chronic or recurrent infectious diseases, or systemic infection caused by fungal, parasitic or mycotic pathogens, or other opportunistic infections;
6. History of active or latent tuberculosis (TB), or inadequately treated latent TB infection, or contact history of patients with TB;
7. Has serious bone or joint infection within 6 months before screening, serious infection (e.g., hospitalization for infection or parenteral antibiotic treatment for infection), or herpes zoster virus infection within 3 months before screening;
8. Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), or treponema pallidum antibody (TP-Ab);
9. Subject with any acute infection, or any symptoms or signs of infection;
10. Has presence of a surgical site, trauma site, severe mucosal ulceration, or incomplete fracture healing, or risk of gastrointestinal bleeding/perforation (e.g., active gastroduodenal ulcer, intestinal obstruction, ulcerative colitis, esophagogastric varices, gastrointestinal perforation within 6 months prior to screening), and risk of infection as assessed by the investigator;
11. Abnormal liver function within 3 months prior to administration, or higher than the upper limit of normal ALT, AST, ALP, or TBL detected during screening period, and is clinically significant;
12. Has abnormal coagulation parameters (including prothrombin time and international normalized ratio) and is clinically significant;
13. Known or suspected history of drug abuse (e.g., morphine, methamphetamine, ketamine, dimethylene dioxyamphetamine, THC, cocaine, etc.), or positive at baseline screening for drug abuse;
14. Alcohol abuse within 1 year prior to screening (drinking more than 14 standard units per week, with 1 standard unit containing 14g of alcohol, such as 360 ml of 5% beer, 45ml of 40% liquor, 120 ml of 12% wine), or positive breath test for alcohol during screening/baseline period;
15. Smokes more than 5 cigarettes per day or the equivalent of 5 cigarettes per day of nicotine-containing products within 3 months before screening, or inability to comply with the smoking ban during the study;
16. Has received vaccines within 3 months prior to screening, or plan to receive vaccines during the study;
17. Has received any experimental drug or participated in any drug/investigational device trial within 3 months before dosing;
18. Has undergone any surgery in the 3 months prior to screening, or planned to undergo surgery during the study period;
19. Subject with previous severe or current chronic diseases of the central nervous system, cardiovascular, liver, kidney, lung, digestive tract, metabolic, hematological, skeletal, immune and other systems of clinical significance, or any other diseases or medical conditions that may affect the study or pose an unacceptable risk to the subject in the judgment of the investigator;
20. History of abdominal surgery affecting the structure and function of the digestive tract;
21. Subject with structural abnormalities of the digestive tract, or previous history of gastrointestinal disease (such as gastrointestinal bleeding, gastrointestinal perforation, gastroesophageal reflux disease, and inflammatory bowel disease) or current clinically significant gastrointestinal disease (such as gallstones) or symptoms (such as nausea, vomiting, and diarrhea), or patients who had undergone gastrointestinal surgery;
22. Subject with symptoms of uninduced diarrhea within 3 months prior to screening;
23. Any clinically significant abnormal results in vital signs, physical examination, or protocol-specified laboratory tests;
24. Any clinically significant abnormal result in 12-lead ECGs, such as QTcF interval (Fridericia correction) > 450 ms for males and > 470 ms for females;
25. Serum creatinine clearance (Ccr) < 90 mL/min, calculated according to Cockcroft-Gault formula: Creatinine clearance (mL/min) =(140-age) × body weight (kg) ×(0.85 [women only])/ 72 × serum creatinine (mg/dL), Or creatinine clearance (mL/min) =(140-age) × body weight (kg) ×(0.85 [women only])/ 0.81 × serum creatinine (μmol/L);
26. Has received any drugs that may interact with the investigational drug within 7 days before administration, such as CYP3A4 inhibitors and inducers, or P-gp inhibitors (refer to Appendix 12.6 for details);
27. Has received any drugs that inhibit or induce hepatic drug-metabolizing enzymes within 7 days before screening; Ingestion of foods or beverages that induce or inhibit liver metabolism enzymes (e.g., grapefruit, etc.) within 48 hours before administration; Inability to comply with the prohibition of ingestion of any foods or beverages containing or metabolically producing caffeine or xanthine (e.g., coffee, tea, chocolate) within 48 hours before the first administration until the completion of the last PK blood sample;
28. Inability to comply with the prohibition of the use of any medications, other than those permitted by the investigator, including prescription and over-the-counter medications (excluding topical eye/nose drops and creams without systemic exposure risk), vitamins (excluding conventional vitamins), health supplements, or Chinese herbal medicine within 14 days or 5 half-lives (whichever is longer) before administration until the last visit.
29. Has donated or lost ≥400 ml of blood within the 3 months prior to screening, or planned to donate blood during the study period;
30. Inability to be venipunctured for blood collection and/or has a history of fainting blood and fainting needles; Subject with any other serious systemic diseases, significant laboratory or procedure abnormalities, or other reasons that, in the opinion of the Investigator, might place the subject at unacceptable risk for participation in this study.

For Psoriasis Patient:

Inclusion Criteria

1. Men and women aged 18-70 at the time of screening visit;
2. Body mass index (BMI) 18-35 kg/m2, inclusive, and total body weight ≥ 40 kg;
3. Patients with plaque psoriasis who meet the following criteria during screening:

   1. Diagnosis of plaque psoriasis for at least 6 months before the first administration, and, in the opinion of the Investigator, have stable psoriasis with no significant progression or morphological changes.
   2. Psoriasis Area and Severity Index (PASI) score 12
   3. Static physician's global assessment (sPGA) ≥3
   4. Psoriatic plaques must cover 10% of body surface area (BSA)
   5. Deemed by Investigator to be eligible for phototherapy or systemic therapy
   6. Subject is willing to discontinue topical and/or systemic therapies other than the investigational drugs, with the exception of topical moisturizer and low-intensity topical steroids used for salvage therapy.
4. Voluntarily participate in the study and provide the signed and dated informed consent；
5. For female subjects:

   1. With no childbearing potential, including those who has surgical sterilization (documented tubal ligation, hysterectomy, or bilateral oophorectomy) at least 6 weeks before the screening visit, and who menopause ≥12 months before the screening visit (confirmed by a follicle stimulating hormone (FSH) level ≥40IU/L), or
   2. With childbearing potential (WOCBP), must not be pregnant nor lactating, and must have used nonpharmacologic contraception 30 days before administration, during the study, and for 3 months after dose, and must have tested negative for human chorionic gonadotropin (hCG) at the screening visit and D-1; female subjects must refrain from egg donation during this period;
6. Males who are sexually active with WOCBP must have used nonpharmacologic contraception 14 days before administration, during the study, and for 3 months after administration. Male subjects must refrain from sperm donation during this time;
7. Subject is willing to comply with protocol-specified visits, treatments, laboratory tests, and other study-related procedures and requirements.

Exclusion Criteria

1. Allergy to the investigational drugs or the excipients, or a history of severe allergy (including any food allergy or drug allergy);
2. Has received IL-17 small molecule inhibitors in the past;
3. Diagnosis of non-plaque psoriasis (guttate, inverse, pustular, erythrodermic);
4. Diagnosis of or at risk for drug-induced psoriasis (including, but not limited to, new-onset psoriasis or exacerbation of psoriasis caused by β receptor blockers, calcium channel inhibitors, or lithium, and newly use of β receptor blockers or calcium channel inhibitors within 2 years prior to enrollment);
5. Has or suspected to have other skin or systemic autoimmune diseases other than psoriasis and psoriatic arthritis;
6. History of lack of response to Ustekinumab, Guselkumab, Tildrakizumab, Secukinumab, Ixekizumab, or Brodalumab (any therapeutic agent targeted to IL-12, IL-17 or IL-23) at approved doses after at least 3 months of therapy;
7. Has received Ustekinumab, Guselkumab, Tildrakizumab, Secukinumab, Ixekizumab, or Brodalumab (any therapeutic agent targeted to IL-12, IL-17 or IL-23) within 3 months of first administration of investigational drugs;
8. Has received TNF-α inhibitor(s) (Etanercept, Infliximab, Adalimumab, or Sacituzumab) within 2 months of first administration of investigational drugs;
9. Has received phototherapy or any systemic medications/treatments for psoriasis, (including, but not limited to, Chinese medicines, JAK inhibitors, PDE4 inhibitors, TYK2 inhibitors, methotrexate, cyclosporin, retinoids) within 1 month of the first administration;
10. Has used topical medications/treatments for psoriasis (including, but not limited to, glucocorticoids, vitamin D derivatives, retinoids, calcineurin inhibitors, aryl hydrocarbon receptor agonists, combination preparation for external use, Chinese medicines, JAK inhibitors, PDE4 inhibitors) within 2 weeks of the first administration;
11. Has received any other monoclonal antibodies that the Investigator determined could affect the evaluation of the investigational drugs. For example, has received natalizumab, efalizumab, or agents that modulate B cells or T cells (eg, alemtuzumab, abatacept, alefacept, or visilizumab) within 3 months of the first administration; or has received rituximab within 6 months of the first administration;
12. Medical history or family history of psychiatric disorders or genetic immunodeficiency;
13. Has received hematopoietic stem cell transplantation, or organ transplantation in the past;
14. History of chronic or recurrent infectious diseases, or systemic infection caused by fungal, parasitic or mycotic pathogens, or other opportunistic infections;
15. History of active or latent TB, or inadequately treated latent TB infection, or contact history of patients with TB;
16. Has serious bone or joint infection within 6 months before screening, serious infection (e.g., hospitalization for infection or parenteral antibiotic treatment for infection), or herpes zoster virus infection within 3 months before screening;
17. Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), or treponema pallidum antibody (TP-Ab);
18. Subject with any acute infection, or any symptoms or signs of infection;
19. Has presence of a surgical site, trauma site, severe mucosal ulceration, or incomplete fracture healing, or risk of gastrointestinal bleeding/perforation (e.g., active gastroduodenal ulcer, intestinal obstruction, ulcerative colitis, esophagogastric varices, gastrointestinal perforation within 6 months prior to screening), and risk of infection as assessed by the Investigator;
20. History of malignant tumor or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell or squamous cell carcinoma, or carcinoma in situ of cervix that has been treated with no evidence of recurrence within the previous 3 years);
21. Class III or IV congestive heart failure by New York Heart Association Criteria; Or has unstable cardiovascular disease, defined as a recent clinical deterioration (e.g., unstable angina, rapid atrial fibrillation) in the last 3 months or a cardiac hospitalization within the last 3 months;
22. Absolute WBC count, lymphocyte count, or neutrophil count is below the lower limit of normal and is clinically significant;
23. Abnormal liver function within 3 months before the first administration, or higher than the upper limit of normal ALT, AST, ALP, or TBL detected during screening period, and is clinically significant；
24. Serum creatinine clearance (Ccr) < 60 mL/min, calculated according to Cockcroft-Gault formula;
25. Has abnormal coagulation parameters (including prothrombin time and international normalized ratio) and is clinically significant;
26. Known or suspected history of drug abuse (e.g., morphine, methamphetamine, ketamine, dimethylene dioxyamphetamine, THC, cocaine, etc.), or positive at baseline screening for drug abuse;
27. Alcohol abuse within 1 year prior to screening (drinking more than 14 standard units per week, with 1 standard unit containing 14g of alcohol, such as 360 ml of 5% beer, 45ml of 40% liquor, 120 ml of 12% wine), or positive breath test for alcohol during screening/baseline period;
28. Smokes more than 5 cigarettes per day or the equivalent of 5 cigarettes per day of nicotine-containing products within 3 months before screening, or inability to comply with the smoking ban during the study;
29. Has received vaccines within 3 months prior to screening, or plan to receive vaccines during the study;
30. Has received an experimental antibody or biologic therapy within the previous 6 months, or received any other experimental therapy or new investigational agent within 30 days or 5 half-lives (whichever is longer) of any study medication administration;
31. Has undergone any surgery in the 3 months prior to screening, or planned to undergo surgery during the study period;
32. Has donated or lost ≥400 ml of blood within the 3 months prior to screening, or planned to donate blood during the study period;
33. Inability to be venipunctured for blood collection and/or has a history of fainting blood and fainting needles;
34. Subject with any other serious systemic diseases, significant laboratory or procedure abnormalities, or other reasons that, in the opinion of the Investigator, might place the subject at unacceptable risk for participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | up to 56 days
Number of participants with clinically significant changes from baseline in vital signs | up to 56 days
Number of participants with clinically significant changes from baseline in clinical laboratory values | up to 56 days
  Safety and tolerability outcome measures include, but are not limited to vital signs, physical examination, 12-lead ECGs, clinical laboratory tests, and adverse events.
Number of participants with clinically significant changes from baseline in physical examination | up to 56 days
Number of participants with clinically significant changes from baseline in 12-lead electrocardiograms(ECGs) | up to 56 days

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to end of dosing interval (AUCtau) for Parts A, B, C and D | up to 72 hours after the last dose
Area under the plasma concentration-time curve from time zero to infinity (AUCinf) for Parts A, B, C, and D | up to 72 hours after the last dose
Maximum observed plasma concentration (Cmax) for Parts A, B, C and D | up to 72 hours after the last dose
Time to maximum plasma concentration (Tmax) for Parts A, B, C and D | up to 72 hours after the last dose
Apparent terminal elimination half-life (t½) for Parts A, B, C and D | up to 72 hours after the last dose
Apparent systemic clearance (CL/F) for Parts A, B, and C | up to 72 hours after the last dose
Apparent volume of distribution (Vz/F) for Parts A, B, and C | up to 72 hours after the last dose
MRT（Mean Residence Time）for Parts A, B, C and D | up to 72 hours after the last dose
Accumulation ratios (Rac) for Parts B and D | up to 72 hours after the last dose
degree of fluctuation（DF）for Parts B and D | up to 72 hours after the last dose
the change in serum IL-17A level from the baseline for Parts A, B and D | up to 72 hours after the last dose
the changes in serum beta-defensin 2(BD-2) from the baseline for Part D | up to 72 hours after the last dose
the changes in serum IL-19 level from the baseline for Part D | up to 72 hours after the last dose
The percentage change in psoriasis area and severity index (PASI) score from the baseline for Part D | up to 56 days
Number of Participants Achieving 50% Improvement from Baseline in PASI (PASI-50) Score for Part D | up to 56 days
Number of Participants Achieving 75% Improvement from Baseline in PASI (PASI-75) Score | up to 56 days
Number of Participants Achieving 90% Improvement from Baseline in PASI (PASI-90) Score | up to 56 days
Number of Participants Achieving a Static Physician's Global Assessment (sPGA) of Clear (0) or Almost Clear (1) for Part D | up to 56 days
The change in sPGA score from the baseline for Part D | up to 56 days
The change in body surface area(BSA) from the baseline for Part D | up to 56 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China